CLINICAL TRIAL: NCT05563298
Title: A Pilot Study Evaluating the Feasibility, Safety, and Efficacy of the Vielight Neuro RX Gamma for the Treatment of Amnestic Mild Cognitive Impairment (aMCI)
Brief Title: Neuro RX Gamma for Amnestic Mild Cognitive Impairment (aMCI)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Corinne Fischer, Professor of Psychiatry, University of Toronto, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 22-128
Record Dates: First submitted 2022-09-16; First posted 2022-10-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: MCI; Amnestic Mild Cognitive Disorder
Keywords: MCI; Photobiomodulation; PBM; AD

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind trial. The trial will include patients with amnestic MCI who will be randomized in a 1:1 ratio to treatment with an active or sham Neuro RX Gamma device.
Who Masked: Participant
Masking Description: This is a randomized, single-blind trial. The trial will include patients with amnestic MCI who will be randomized in a 1:1 ratio to treatment with an active or sham Neuro RX Gamma device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Neuro Rx Device (Active Comparator): The active device will deliver light for the 20 minutes session duration.
  Interventions: Device: Neuro RX Gamma device
- Sham Neuro Rx Device (Sham Comparator): The Sham device is indistinguishable from the active device. The sham device will not deliver light for the 20 minutes session duration.
  Interventions: Device: Sham Neuro RX Gamma device

INTERVENTIONS:
Device: Neuro RX Gamma device — The Neuro RX Gamma device is a portable, wearable, low level light therapy (LLLT) delivery device. The Vielight Neuro RX Gamma delivers a synchronized pulse frequency of 40 Hz from all LED clusters.
  Arms: Active Neuro Rx Device
Device: Sham Neuro RX Gamma device — The Sham device is indistinguishable from the active device. The sham device will not deliver light for the 20 minutes session duration.
  Arms: Sham Neuro Rx Device

SUMMARY:
Over 50 million people worldwide are currently living with dementia-a number projected to rise to 152 million by 2050. Mitochondrial dysfunction in the brains of individuals with Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD) has gained increasing attention as a potential mechanism and therapeutic target. However, no effective treatment specifically targeting mitochondrial function is currently available.

Photobiomodulation (PBM) is an innovative, non-invasive technique that delivers near-infrared light transcranially to the brain. PBM is believed to enhance mitochondrial function-particularly in tissues with high mitochondrial density such as the brain-by reducing oxidative stress and increasing ATP production. It can be safely administered to awake outpatients and does not require general anesthesia or surgical intervention. While preclinical and case studies suggest PBM may be beneficial in AD, the absence of placebo-controlled trials and objective biomarkers has limited understanding of its effectiveness and underlying mechanisms.

Objectives: This pilot feasibility study aims to assess cognitive outcomes and neural correlates associated with PBM in individuals with early amnestic MCI (aMCI). Participants who meet eligibility criteria (n = 20) will undergo a 6-week, home-based PBM intervention using the Neuro Rx Gamma device (6 days/week, 20 minutes/session). Clinical and cognitive assessments, blood sample collection, and structural and resting-state functional MRI scans will be conducted at two time points: baseline and post-treatment. These assessments will enable evaluation of PBM's effects on cognition and brain function, with particular focus on mitochondrial-related mechanisms.

This study offers a unique opportunity to investigate whether PBM can modulate mitochondrial and neural processes associated with cognitive decline in aMCI.

DETAILED DESCRIPTION:
Intervention:

The experimental intervention will be the Vielight Neuro RX Gamma photobiomodulation (PBM) device, which delivers near-infrared light via five light-emitting diodes (LEDs) operating at a wavelength of 810 nm. The LEDs are positioned equidistantly on the scalp and intranasally to target key brain regions. The device generates no significant heat, enabling the use of an indistinguishable sham device for placebo control.

All participants will self-administer 20-minute sessions once daily, six days per week, for six weeks. Subjects and/or caregivers will receive training to ensure proper at-home use and will be asked to maintain a treatment diary to monitor adherence.

Assessments:

Each participant will undergo two in-person visits-at baseline (T0) and post-intervention (week 7; T2)-to complete the following evaluations:

Mini-Mental State Examination (MMSE) California Verbal Learning Test - Long Delayed Free Recall (CVLT-LDFR) Trail Making Test A and B (TMT-A, TMT-B)

Pittsburgh Sleep Quality Index (PSQI) Mild Behavioral Impairment Checklist (MBI-C) Blood tests: lactate and lactate-to-pyruvate (L/P) ratio Structural and resting-state functional MRI, 1H-MRS, CBF An additional safety check will be conducted at week 1, 3, 5, and at the end of the study (either remotely or in person).

Safety Endpoints:

Serious adverse events (SAEs), regardless of device causality Device-related adverse events (AEs) Rates of epistaxis (nosebleeds) and nasal infections

ELIGIBILITY:
Inclusion Criteria:

* Age is greater than or equal to 50 years old.
* Meets the National Institute on Aging and Alzheimer's Association (NIA-AA) criteria for MCI due to Alzheimer's disease.
* Essentially normal functional activities as derived from the CDR.
* If receiving ongoing cholinesterase inhibitor therapy and/or memantine, must be on a stable dosage for at least the prior 3 months.
* MoCA score between 19 and 25 at screening assessment and impairment in learning and memory domain.

Exclusion Criteria:

* Cannot tolerate blood draws.
* Claustrophobia (fear of small or enclosed spaces), that cannot tolerate MRI scanners.
* A pace-maker or other metal implants that would preclude safe use of MRI.
* DSM 5 diagnosis of alcohol or other substance use disorders within the past 12 months.
* Unstable medical illness, (e.g., uncontrolled diabetes mellitus or hypertension).
* Any history of stroke, seizures, MS, light sensitivity or Lyme disease.
* Any issues with ambulation, vision, or hearing which could, in the opinion of the investigator, interfere with their ability to complete assessments.
* Participant or caregiver does not speak English at a level necessary for the completion of the assessments.
* Has not completed at least a grade eight education, as necessary for the completion of the assessments.
* Currently participating in another clinical research study involving an investigational product.
* History of significant agitation and/or aggression, epileptic seizures.
* Current neurologic disease affecting cognition other than Alzheimer's disease.
* Photosensitivity reactions to sunlight or visible light (polymorphous light eruption, solar urticaria, persistent light reactivity).
* History of recurrent epistaxis within the last 24 weeks or currently taking major anti-coagulants (including warfarin, low molecular weight heparin)
* Increased skin sensitivity at the treatment site including active herpes simplex in the treatment area, history of keloid formation, or history of retinoid use in the past month.
* Pregnant or lactating or planning to become pregnant.
* Currently undergoing light therapy treatment.
* Any reason that, in the opinion of the investigator, might place a participant at unacceptable risk for participation in the trial.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Changes from pre- to post-treatment on mental status and cognitive function assessed by Mini-Mental State Examination (MMSE) | Assessed at baseline and post-intervention (week 7)
  MMSE is a brief 30-point assessment
Changes from pre- to post-treatment on verbal learning and memory assessed by California Verbal Learning Test-II (CVLT-II) | Assessed at baseline and post-intervention (week 7)
  The Composite Score was created by grouping variables into domains and averaging the domains into a single Composite Score for each participant using:
  CVLT-II - Total Recall Trials 1-5 CVLT-II - d' Hits and False Alarms of recognition Yes/No responses CVLT-II - Percent retained at long delay trial from trial 5 at immediate recall condition
Changes from pre- to post-treatment on processing speed assessed by Trail Making Test (TMT)-part A & B | Assessed at baseline and post-intervention (week 7)
  Trail Making A - Time per correct connection

SECONDARY OUTCOMES:
Changes from pre- to post-treatment on peripheral blood-biomarkers assessed by blood | Assessed at baseline and post-intervention (week 7)
  Blood lactate and lactate/pyruvate ratio will be measured due to their noted relationship with mitochondrial function.
Changes from pre- to post-treatment on plasma biomarkers | Assessed at baseline and post-intervention (week 7)
  markers of neuroinflammation (IL-6, IL-10), neurodegeneration (GFAP, NfL), tau pathology (phosphorylated Tau-217), and synaptic plasticity (Brain-Derived Neurotrophic Factor-BDNF)
Changes from pre- to post-treatment on Neuropsychiatric symptoms (NPS) using MBI-C (Mild Behavioral Impairment Checklist) | Assessed at baseline and post-intervention (week 7)
  The MBI-C is a 34-item instrument and serves as a global and domain-specific NPS measure including early symptom presentations
Changes from pre- to post-treatment on structural MRI (T1-weighted imaging) | Assessed at baseline and post-intervention (week 7)
  Cortical thickness and subcortical volume
Changes from pre- to post-treatment on brain metabolites (PCC) | Assessed at baseline and post-intervention (week 7)
  N-acetylaspartate/creatine, lactate/creatine via single-voxel ¹H-MRS
Changes from pre- to post-treatment on structural MRI (Diffusion tensor imaging - DTI) | Assessed at baseline and post-intervention (week 7)
  fractional anisotropy (FA), and mean diffusivity (MD) measure
Changes from pre- to post-treatment on resting state functional connectivity of the default mode network (DMN) via rs-fMRI | Assessed at baseline and post-intervention (week 7)
  Brain networks functional connectivity
Changes from pre- to post-treatment on Pittsburgh sleep quality index | Assessed at baseline and post-intervention (week 7)
  The measure consists of 19 individual items, creating 7 components that produce one global score
Changes from pre- to post-treatment on cerebral blood flow (CBF) | Assessed at baseline and post-intervention (week 7)
  CBF using pseudo-continuous arterial spin labeling (PCASL) -with a focus on DMN

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Fischer, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No